CLINICAL TRIAL: NCT03898037
Title: Effect of Lifestyle and/or Metformin Intervention on Pregnancy Outcome in Overweight/Obese Non-pcos Infertility Women With Insulin Resistance , A Pilot Randomized Controlled Trial
Brief Title: Effect of Lifestyle and/or Metformin Intervention on Pregnancy Outcome, A Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P2019001
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Infertility, Female; Obesity; Insulin Resistance
MeSH Terms: conditions — Infertility, Female; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lifestyle intervention group (Experimental): Subjects will receive weight loss intervention under the guidance of a dietitian after assigned to lifestyle intervention group, including: restricted energy balanced diet, aerobic exercise, etc. Subjects will come to the hospital to measure their height, weight, waist circumference, hip circumference, body fat rate, BMI and test oral glucose tolerance test (OGTT)/insulin resistance test(IRT)/HOMA, blood routine, liver and kidney function on the day of grouping and in the 4th week, the 8th week, the 12th week after grouping.
  The aim is to lose 5-10% of the initial body weight. If the target was reached within 3 months, subjects will receive ovarian stimulation treatment in advance, otherwise treatment starts after 3 months. All subjects are treated with the same procedures，including a long ovarian stimulation regimen, oocyte retrieval, and fertilization, followed by a planned transfer of two day-3 embryos. The pregnancy and perinatal outcomes after transfer were followed up.
  Interventions: Behavioral: weight loss intervention
- metformin intervention group (Experimental): Subjects will be given metformin intervention with a starting dose of 0.5g bid after assigned to metformin intervention group, and the dose will be adjusted by doctors according to the insulin level and adverse events. Subjects will come to the hospital to measure their height, weight, waist circumference, hip circumference, body fat rate, BMI and test OGTT/IRT/HOMA, blood routine, liver and kidney function on the day of grouping and the 4th week, the 8th week, the 12th week after grouping.
  The aim is to adjust insulin level to normal within 3 months. If the target was reached within 3 months, subjects will start to receive ovarian stimulation treatment in advance, Otherwise treatment starts after 3 months. All subjects are treated with the same procedures, including a long ovarian stimulation regimen, oocyte retrieval, and fertilization, followed by a planned transfer of two day-3 embryos etc. The pregnancy and perinatal outcomes after transfer were followed up.
  Interventions: Drug: metformin intervention
- lifestyle combined with metformin intervention group (Experimental): Subjects will receive weight loss intervention and metformin intervention after assigned to lifestyle combined with metformin intervention group. Subjects will come to the hospital to measure their height, weight, waist circumference, hip circumference, body fat rate, BMI and test OGTT/IRT/HOMA, blood routine, liver and kidney function on the day of grouping and in the 4th week, the 8th week, the 12th week after grouping.
  The aim is to lose 5-10% of the initial body weight and adjust insulin level to normal within 3 months. If the target was reached within 3 months, subjects will receive ovarian stimulation treatment in advance, otherwise treatment starts after 3 months. All subjects are treated with the same procedures，including a long ovarian stimulation regimen, oocyte retrieval, and fertilization, followed by a planned transfer of two day-3 embryos etc. The pregnancy and perinatal outcomes after transfer were followed up.
  Interventions: Behavioral: weight loss intervention; Drug: metformin intervention
- routine clinical education group (No Intervention): Subjects will only accept clinical routine education after assigned to routine clinical education group. Subjects will measure their height, weight, waist circumference, hip circumference, body fat rate, BMI and test OGTT/IRT/HOMA, blood routine, liver and kidney function on the day of grouping and will start induced ovulation therapy after completing routine clinical examination. All subjects are treated with the same procedures，including a long ovarian stimulation regimen, oocyte retrieval, and fertilization, followed by a planned transfer of two day-3 embryos etc. The pregnancy and perinatal outcomes after transfer were followed up.

INTERVENTIONS:
Behavioral: weight loss intervention — weight loss intervention under the guidance of a dietitian, including: restricted energy balanced diet, aerobic exercise, etc.
  Arms: lifestyle combined with metformin intervention group; lifestyle intervention group
Drug: metformin intervention — metformin intervention with a starting dose of 0.5g bid, and the dose will be adjusted by doctors according to the patient's insulin level and adverse events.
  Arms: lifestyle combined with metformin intervention group; metformin intervention group

SUMMARY:
The purpose of pilot trial is to compare the efficacy of lifestyle intervention, metformin intervention, lifestyle combined with metformin intervention in improving assisted reproductive technology in non-polycystic ovary syndrome(pcos) patients with overweight/obesity and insulin resistance compared with conventional clinical education. Subjects who meet the inclusion criteria will be randomized to four groups: lifestyle intervention group, metformin intervention group, lifestyle combined with metformin intervention group, and routine clinical education group. Subjects of above three intervention group will start ovulation stimulation treatment after reach the aim or duration of intervention and routine clinical education group has no intervention. All subjects are treated with the same procedures, including a long ovarian stimulation regimen, oocyte retrieval, and fertilization, followed by a planned transfer of two day-3 embryos. The primary outcome is ongoing pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 18 to 36 years.
2. Women BMI at least 25kg/m2.
3. Women who are non-pcos patient(2003 Rotterdam criteria).
4. Women with insulin resistance (HOMA criteria).
5. Women who are participating in their first or second fresh embryo cycle of in- vitro fertilization(IVF) or intracytoplasmic sperm injection (ICSI).
6. Women who are indicated IVF or ICSI.

Exclusion Criteria:

1. Women with endometriosis.
2. Women with untreated hydrosalpinx.
3. Women with a uterine cavity abnormality, such as a uterine congenital malformation; untreated uterine septum(except shallow uterine septum), adenomyosis, submucous myoma, or intrauterine adhesions.
4. Women who are indicated and planned to undergo preimplantation genetic diagnosis(PGD)/preimplantation genetic screening(PGS).
5. Women with endocrine abnormalities, such as Cushing syndrome, congenital adrenal hyperplasia, pituitary amenorrhea, thyroid dysfunction etc.
6. Women who had participated in other treatments known to affect diet or weight (such as diet drugs and dietitian intervention) for past 3 months.
7. Women who are unable to follow verbal and written instructions.
8. Women who use donated oocytes to achieve pregnancy.
9. Women with poor ovarian response(Bologna criteria).
10. Women with diabetes mellitus, abnormal glycosylated hemoglobin.
11. Women who has a history of recurrent spontaneous abortion.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
recruitment rate | 10 months
  the proportion of eligible patients randomised

SECONDARY OUTCOMES:
mean numbers of randomised participants per month | 10 months
  numbers of randomised participants / the duration of recruitment
the proportion of participants with good intervention compliance | 16 months
  numbers of participants with good intervention compliance / numbers of participants who received the intervention
the proportion of participants who crossed over from one allocated group to the other | 16 months
  numbers of participants who crossed over from one allocated group to the other / numbers of participants who received the intervention
Proportion of subjects who initiated infertility treatment according to the schedule | 16 months
  numbers of participants who initiated infertility treatment according to the schedule/ numbers of participants who received the intervention
the proportion of participants who completed follow-up | 26 months
  numbers of participants who completed follow-up/ numbers of participants who received the intervention
Biochemical Pregnancy Rate | 16 months
  Number of women with Biochemical pregnancy /number of women who received the intervention Biochemical pregnancy was defined as a human chorionic gonadotropin level of more than 10 milli-International unit（mIU）per milliliter（ml）, as measured at about 14 days after embryo transfer.
Clinical Pregnancy Rate | 18 months
  Number of women with clinical pregnancies /number of women who received the intervention. Clinical pregnancy was defined as the presence of a gestational sac in the uterine cavity at about 28 days after embryo transfer, as detected on ultrasonography.
Live Birth Rate | 26 months
  Numbers of Live birth /number of women who received the intervention.Live birth defined as the delivery of any viable infant at 28 weeks or more of gestation.
Birth weight | 26 months
  Weight of newborns at delivery.
Pregnancy Loss Rate | 26 months
  Number of pregnancy losses / number of clinical pregnancies. Pregnancy loss refers to a complete spontaneous abortion or a nonviable pregnancy before 28 weeks of gestation.
Incidence of moderate to severe ovarian hyperstimulation syndrome(OHSS) | 16 months
  Number of cycles of moderate to severe OHSS/total number of fresh stimulation cycle.
Cumulative incidence of maternal and neonatal complications during whole gestation and prenatal stage | 26 months
  Number of pregnancies with complications / number of pregnancies; Number of live births with neonatal complications / number of live births；

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China

REFERENCES:
- [Derived] Wang X, Cai S, Tang S, Yang L, Tan J, Sun X, Gong F. Effect of lifestyle or metformin interventions before IVF/ICSI treatment on infertile women with overweight/obese and insulin resistance: a factorial design randomised controlled pilot trial. Pilot Feasibility Stud. 2023 Sep 12;9(1):160. doi: 10.1186/s40814-023-01388-x. PMID 37700375